CLINICAL TRIAL: NCT01445366
Title: Solute Removal With High Volume Hemodiafiltration Versus Long High Flux Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011/591
Record Dates: First submitted 2011-09-22; First posted 2011-10-03 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with end-stage renal disease (Experimental)
  Interventions: Device: High volume post dilution hemodiafiltration; Device: high flux hemodialysis

INTERVENTIONS:
Device: High volume post dilution hemodiafiltration — The midweek dialysis sessions of the patients is changed once to a 4 hours high volume post dilution hemodiafiltration (HDF) session, and once to an 8 hours high flux hemodialysis (HD) session.
Device: high flux hemodialysis — The midweek dialysis sessions of the patients is changed once to a 4 hours high volume post dilution hemodiafiltration (HDF) session, and once to an 8 hours high flux hemodialysis (HD) session.

SUMMARY:
This is a prospective cross-over study including 10 stable hemodialysis patients with chronic kidney disease stage 5. The cross-over study lasts 2 weeks with the study dialysis sessions at midweek.

During one session, the patient will be dialyzed during 4 hours with high volume post dilution hemodiafiltration (HDF) with an FX800 hemodialyzer (Fresenius Medical Care) and a blood flow of 300mL/min, dialysate flow of 500mL/min, and substitution flow of 75mL/min.

During the other midweek session, the patient will be dialyzed during 8 hours with high flux hemodialysis (HD) with an FX80 hemodialyzer (Fresenius Medical Care) and a blood flow of 200mL/min and a dialysate flow of 500mL/min.

The HDF and HD sessions will be randomized. Blood samples will be drawn pre and post dialysis from the arterial blood line, and after 30min after dialysis start, a blood sample will be drawn from the inlet and outlet line.

At the dialysate outlet line, partial dialysate collection is performed at the outlet line.

Blood and dialysate samples will be analyzed for a broad range of retention solutes like small and water soluble solutes, middle molecules, and protein bound solutes.

These data will be further used to calculate solute removal and evaluate any differences between the solute removal during high volume post dilution HDF and high flux HD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (CKD) stage 5 with hemodialysis or hemodiafiltration treatment for more than three months.
* No vascular access related problems (Arteriovenous (A/V) fistula, graft or bi-flow catheter)
* Double needle/lumen vascular access
* No ongoing infection
* Singed informed consent form

Exclusion Criteria:

* Inclusion criteria not met
* Known HIV or active hepatitis B or C infection (Positive Polymerisation Chain Reaction (PCR))
* Pregnancy
* Unstable clinical condition (e.g. cardiac or vascular instability)
* Known coagulation problems
* Patients participating in another study interfering with the planned study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2014-09-29 (Actual); Study Completion 2014-09-29 (Actual)

PRIMARY OUTCOMES:
Uremic retention solute concentrations from pre and post dialysis blood samples,dialyzer inlet and outlet blood samples,and spent dialysate samples. | During 4 hours
  Blood and dialysate samples will be analyzed for the concentration of small water soluble solutes, protein bound solutes and middle molecules. Concentrations will be used to calculate different adequacy parameters in order to compare HDF with hemodialysis (HD). Pre to post dialysis during 4h post dilution hemodiafiltration (HDF).
Uremic retention solute concentrations from pre and post dialysis blood samples,dialyzer inlet and outlet blood samples,and spent dialysate samples. | During 8 hours
  Blood and dialysate samples will be analyzed for the concentration of small water soluble solutes, protein bound solutes and middle molecules. Concentrations will be used to calculate different adequacy parameters in order to compare HDF with HD. Pre to post dialysis during 8h high flux HD.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be